CLINICAL TRIAL: NCT05785949
Title: A Prospective, Multicenter, Randomized, Parallel Controlled Study Evaluating the Safety and Efficacy of Chondro-Gide® Bilayer Collagen Membrane in Knee Cartilage Defect Repair
Brief Title: Chondro-Gide® Bilayer Collagen Membrane in Knee Cartilage Defect Repair
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Geistlich Pharma AG (Industry)
Collaborators: TigerMed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13575-238
Record Dates: First submitted 2023-02-14; First posted 2023-03-27 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Cartilage Defects
Keywords: Chondro-Gide®
MeSH Terms: interventions — Arthroplasty, Subchondral

STUDY DESIGN:
Intervention Model Description: In this study, parallel-controlled design is adopted. The experimental group and the control group will complete the study under the same study conditions at basically synchronous study time.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessors will be blinded, i.e., the outcome assessors will not participate in the operation and do not know the subject grouping information. The outcome assessors will make efficacy judgment based on MRI results, so as to reduce study bias caused by subjective assessment error.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Microfracture + Chondro-Gide® (Experimental): Microfracture + Chondro-Gide® bilayer collagen membrane
  Interventions: Procedure: Microfracture; Device: Chondro-Gide bilayer collagen membrane
- Microfracture (Active Comparator): Microfracture
  Interventions: Procedure: Microfracture

INTERVENTIONS:
Procedure: Microfracture — Use of standard tool kit to drill vertically from the periphery to the center with a hole spacing of 3~4 mm with care to prevent penetrating adjacent holes. The hole depth should be 3~5 mm and fat droplets or blood oozing is seen after loosening the tourniquet. However, no blood oozing is observed in some holes and in such case, the hole depth should be deepened to 5~7 mm.
Device: Chondro-Gide bilayer collagen membrane — After the Microfracture, the porous layer of the bilayer collagen membrane faces the bone surface. The already trimmed, cut and wetted membrane is insert into the defect and fixed symmetrically with absorbable surgical suture with needle. Knots are put on the pinhole of collagen membrane to avoid tearing of surrounding cartilage or collagen membrane during knotting.
  Arms: Microfracture + Chondro-Gide®

SUMMARY:
A prospective, multicenter, randomized, parallel controlled study evaluating the safety and efficacy of Chondro-Gide® bilayer collagen membrane in knee cartilage defect repair. The objective of this clinical trial is to evaluate the efficacy and safety of Chondro-Gide® bilayer collagen membrane in knee cartilage defect repair

DETAILED DESCRIPTION:
This is a prospective, multicenter, randomized, parallel controlled and superiority clinical trial. It is planned to be carried out in hospitals with qualifications as a national-level clinical trial institution. Subjects who have signed the ICF, meet all inclusion criteria and do not meet any exclusion criteria will be included in this study. Subjects included will be randomly assigned into the experimental group and the control group at a ratio of 1:1. Those in the control group will receive microfracture, and those in the experimental group will receive microfracture plus Chondro-Gide® bilayer collagen membrane. The primary efficacy evaluation indicator of this clinical study is the MOCART score at 24 months postoperative. The secondary efficacy evaluation indicators are IKDC score (before operation, 3, 6, 12 and 24 months postoperative), MOCART score (6 and 12 months postoperative), hyaline cartilage production (T2 mapping ratio) (12 and 24 months postoperative), Lysholm score (before operation, 3, 6, 12 and 24 months postoperative), and device performance evaluation of the investigational product. Safety evaluation indicators include adverse events (or serious adverse events), device-related adverse events (or serious adverse events), device deficiencies and laboratory examination.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 18-55 years (including 18 years and 55 years);
2. Localized cartilage defects on knee joint, the size of the defect after debridement is 2.0 squared cm - 8.0 squared cm (including 2.0 squared cm and 8.0 squared cm), which was classified by the International Cartilage Repair Society (ICRS) as grade Ⅲ or grade IV;
3. The subjects voluntarily consent to participate in this trial and sign the informed consent form (ICF).

Exclusion Criteria:

1. Body mass index (BMI) ≥ 30 kg/meter squared (BMI = weight divided by height squared);
2. Unilateral knee cartilage defect with the ICRS classification of grade III or grade IV, and with three or more defects;
3. Patients with abnormal lower limb mechanical axis requiring correction, except those that could be corrected during the treatment of cartilage injury;
4. Varus or valgus of lower limb axis > 5°, requiring osteotomy for correction;
5. Patients with multiple ligament injury or total meniscectomy;
6. Those who are known to be allergic to porcine-derived materials or collagen, or refuse to use porcine-derived medical products;
7. Those with severe arthroclisis or arthrofibrosis;
8. Those who have received open knee surgery in the past 6 months;
9. Those who have received microfracture, mosaicplasty or autologous cartilage implantation in the past 3 months;
10. Those who have serious primary cardiovascular diseases, lung diseases, endocrine and metabolic diseases (severe diabetes, severe osteoporosis) or serious diseases affecting their survival, and are considered unsuitable for inclusion by the investigators;
11. Pregnant and lactating women, or those who plan to conceive during the trial, and those who have positive blood/urine pregnancy test results before the trial;
12. Patients with knee infection；
13. Those with connective tissue diseases;
14. Those with nervous system diseases or muscle degeneration;
15. Patients who participated in drug clinical trials within 3 months prior to the enrollment or patients who participated in any other device clinical trials within 1 months prior to the enrollment;
16. Other circumstances which are considered by the investigator not suitable for enrollment in this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2023-04-13 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Magnetic Resonance Observation of Cartilage Repair Tissue (MOCART) | 24 months postoperative
  Cartilage repair is evaluated by MOCART score from nine aspects, such as degree of defect repair and filling of the defect, integration to border zone, surface of repair tissue, structure of the repair tissue, adhesions and subchondral lamina.

SECONDARY OUTCOMES:
International Knee Documentation Committee (IKDC) score | before operation and at 3, 6, 12 and 24 months postoperative
  The therapeutic effect for subjects is evaluated based on the difference between IKDC score at the different timepoints. The score ranges from 0 - 87 points, where higher scores mean a better outcome.
Magnetic Resonance Observation of Cartilage Repair Tissue (MOCART) | 6 and 12 months postoperative
  Cartilage repair is evaluated by MOCART score from nine aspects, such as degree of defect repair and filling of the defect, integration to border zone, surface of repair tissue, structure of the repair tissue, adhesions and subchondral lamina. The Score ranges from 0 - 100, where higher scores mean a better outcome.
Hyaline cartilage production (T2 mapping ratio) | 12 and 24 months postoperative
  Please refer to YY/T 1636-2018 Tissue engineering medical device products-In vivo evaluation of knee cartilage implanted tissue using MRI technique for the specific operation, measurement and evaluation method of T2 mapping technology of MRI.
Lysholm score | before operation and at 3, 6, 12 and 24 months postoperative
  The Lysholm score is assessing patient's knee specific symptoms. The total Lysholm score is 100 (0: worst, 100: best).
Device performance evaluation questionnaire | perioperative (after surgical intervention), on the day of surgery
  The investigator evaluates the performance of the device based on a questionnaire. The evaluation criteria are as follows. There are three answer options to every question:
  1. Is the product operation convenient?
  2. Is the product easy to trim?
  3. Is the product easy to fix?
  4. Is the product compliant after being fixed?
Safety indicators; adverse events and device deficiencies | through study completion, an average of 2 years
  1. Incidence (%) and number of (serious) adverse events, and those of device-related (serious) adverse events;
  2. Incidence (%) and number of device deficiencies;
Safety indicators; Laboratory examination | before operation, 7 days and 6 months postoperative
  Determination of clinical significance of laboratory examination: 1) normal; 2) abnormal but without clinical significance; 3) abnormal with clinical significance; 4) not examined. If the clinical significance is judged as 3) abnormal with clinical significance, the abnormality is explained, followed up, and reexamined until normal or reaching baseline level or stable.

CONTACTS AND LOCATIONS:
Overall Officials: Fabiana Martinelli, Study Director — Geistlich Pharma AG
Locations (18):
- China (18):
  - Shen Zhen Secondary People hospital, Shenzhen, Guangdong
  - Peking University Shen Zhen hospital, Shenzhen, Guangdong
  - The Second People Hospital of Yi Bin, Yibin, Guangdong
  - The Second Hospital of Tang Shan, Tangshan, Hebei
  - Nan Chang First Hospital, Nanchang, Jiangxi
  - QiLu Hospital of Shan Dong University, Jinan, Shandong
  - The First People Hospital of Ka Shi, Kashgar, Xinjiang
  - Tai Zhou Hospital of Zhe Jiang Province, Taizhou, Zhejiang
  - Sino-Japanese Friendship Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - The Second Hospital of Jilin University, Changchun
  - The First Affiliated Hospital of Jinan University, Guangzhou
  - The Third Affiliated Hospital of Southern Medical University, Guangzhou
  - The second affiliated hospital of Zhejiang University School of Medicine, Hanzhou
  - Inner Mongolia People's Hospital, Hohhot
  - The First Affiliated Hospital of Kunming Medical University, Kunming
  - The First Affiliated Hospital Of Nanchang University, Nanchang
  - The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School, Nanjing

IPD SHARING:
Plan to Share IPD: No